CLINICAL TRIAL: NCT06166953
Title: The Effect of Digital Technology-Supported Education and Monitoring on Anxiety, Pain, Sleep and Quality of Life in Patients Undergoing Immediate Breast Reconstruction After Mastectomy: A Randomized Controlled Study
Brief Title: The Effect of Digital Technology-Supported Education on Patients Undergoing Breast Reconstruction After Mastectomy: A Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Aylin Günay, MSc, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA22/498
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; mobile application; nursing care; technology; surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A mobile application will be developed by software engineer including informational needs of breast cancer patients starting prior to surgery lasting to discharge. Expert opinion will be obtained about contents of mobile application. The application will be downloaded smart phones of patients for use when needed. Patients who meet the inclusion criteria will be informed about the research by the researcher according to the randomization list, and their consent will be obtained from those who agree to participate in the research. Due to the study design, patients will not know which intervention is being applied to them, and it will be done single-blinded. The application will be carried out by the researcher knowing the patients in the intervention and control groups. The analysis of the data coded as A and B will be done by a statistician.
Who Masked: Participant, Outcomes Assessor
Masking Description: Those who accepted the study were asked to read the "Informed Volunteer Consent Form" indicating that they volunteered to participate in the study, and the control and intervention group patients were instructed not to share information about the application with each other in order to prevent them from being influenced by each other in the outpatient clinic environment/institution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile application (Experimental): The mobile application will be downloaded on smart phones of participants. This group will be able to look up information related to surgical period when needed.
  Interventions: Other: digital technology-supported education
- Control (No Intervention): The control group will receive routine care. This group will wear smart band for pulse rate, sleep, blood pressure, and SpO2 record for data collection times.

INTERVENTIONS:
Other: digital technology-supported education — The education will include information about surgical process and care after surgery.
  Arms: mobile application

SUMMARY:
The goal of this randomized, controlled study is to test the effectiveness of digital technology-supported education on patients undergoing breast reconstruction after mastectomy.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in our country and all over the world, and there are surgery, radiotherapy, chemotherapy, hormonal and targeted treatment options in the treatment of patients diagnosed with breast cancer. Surgery is an important option for the majority of patients diagnosed with breast cancer, and breast-conserving surgery and mastectomy are frequently performed. Patients who undergo mastectomy can also choose breast reconstruction surgeries, which enable the reconstruction of breast tissue through various methods, because they feel better both psychologically and physiologically.

Breast reconstruction can be performed in two periods: early and late. Patients who undergo breast reconstruction simultaneously with mastectomy may experience psychological problems such as anxiety, depression and fear in the preoperative period, and patients may experience surgery-related bleeding, hematoma, seroma, wound infection, tissue necrosis, fat necrosis, capsule contraction, implant loss and pain. Complications may develop and individuals' quality of life may be negatively affected. Patients need support care, treatment and preventive health interventions, and education on late effects/long-term physical and psychosocial problems in order to maintain their independence in daily activities and improve their quality of life.

In addition to written, visual and audio materials in patient education, mobile applications and wearable technologies come to the fore with developing and advancing technology. Mobile health service offered starting from the pre-operative period; In addition to heart rate, blood pressure, oxygen saturation, blood glucose level, daily drainage monitoring, spirometry results and medication compliance; Pain level, sleep quality, daily living activities and exercise level can be evaluated, and the quality of care is increased with nursing care practices and continuity of education.

This study aims to determine the effect of mobile technology-supported education and monitoring on care outcomes in patients who underwent breast reconstruction simultaneously with mastectomy due to breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with stage 1, 2, or 3 breast cancer
* Planned to undergo immediate breast reconstruction after mastectomy for the first time
* Being between 18 to 75 years old
* Able to use smart phone
* Having smart phone with Android v5.0 or iOS v9.0 and above software, Bluetooth and internet connection
* Having no hearing or visual impairment
* Having no physical limitation
* Turkish speaking volunteers

Exclusion Criteria:

* Patients planned to undergo total abdominal hysterectomy and bilateral salpingo oophorectomy with immediate reconstruction after mastectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline and 30th days
  The Hospital Anxiety and Depression Scale will be used. It is a valid and reliable scale in Turkish. The higher score the higher risk for depression or anxiety. (Change from baseline to 5th, 15th and 30th days will be assessed).
Surgical pain | (Change from baseline to 5th, 15th and 30th days will be assessed).
  Visual Analogue Scale (VAS): It is used to evaluate the subjective discomfort states of patients. It consists of a horizontal line 10 cm long. It is a ruler with the left side stating "no pain" and the right side stating "the worst pain" (unbearable pain). Values range from 0 to 10, with higher values indicating increased discomfort. It is easy to apply. It has been shown to be sensitive to pain and discomfort.
Sleep quality | (Change from baseline to 5th, 15th and 30th days will be assessed).
  Pittsburg Sleep Quality Index: It is valid and reliable scale. in Turkish language.The scale consists of 24 questions, 19 of which are feedback questions and 5 of which are to be answered by the spouse or roommate. When calculating the index score, questions answered by the individual's spouse or roommate are not included in the calculation. Self-assessment questions include various items related to sleep quality. These are to determine sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems. The 18 items scored are grouped into 7 component scores. Some of the components consist of a single substance, while others are obtained by grouping several substances. Each item is evaluated with a score between 0-3. The sum of these seven component scores gives the total index score. Total score is between 0-21. A high total score indicates poor sleep quality.
Quality of life after surgery | (Change from baseline to 5th, 15th and 30th days will be assessed).
  SF-12 Quality of Life Scale (SF-12), is a scale that evaluates the quality of life for the last four weeks without focusing on a specific age group or disease group. High scores indicate good health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share IPD .